CLINICAL TRIAL: NCT02248649
Title: A Telemedicine Intervention to Improve Cognitive Function in Patients With PD
Brief Title: Telemedicine Intervention to Improve Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N1696-I
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Exercise therapy; Mild cognitive impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity (Experimental): Structured walking program
  Interventions: Behavioral: Structured physical activity
- Control (Active Comparator): Health education attention control
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Structured physical activity — Walking instruction and encouragement
  Arms: Physical Activity
Behavioral: Health education — Provision of general information about a variety of health topics
  Arms: Control

SUMMARY:
This project is investigating whether a home-based exercise program will reduce cognitive decline in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background/Rationale:

Progressive cognitive impairment leading to dementia is an important component of Parkinson's disease (PD), contributing to significant levels of disability. The number of Veterans who will develop PD and, in turn, the number of Veterans with PD who develop dementia is likely to increase substantially. Given the profound negative health and social consequences associated with the development of dementia, it is critical to identify interventions that effectively slow the decline of cognitive function to prolong the time to onset of dementia. Based on the results of prior studies, physical activity is one of the few nonpharmacological interventions that holds promise in slowing cognitive decline.

Objective:

The investigators hypothesize that a home-based physical activity intervention to promote walking will reduce cognitive decline in Veterans with mild cognitive impairment in PD (PD-MCI).

Methods:

The proposed study is a randomized, controlled trial of a home-based walking intervention, evaluating effects on cognitive function. Community-dwelling Veterans with PD-MCI will be randomized to a walking intervention or a health education control intervention. Subjects will be male and female Veterans with a physician diagnosis of idiopathic, typical PD, with at least 2 of 3 cardinal signs of PD, response to dopaminergic medication, and MCI. The interventions will last 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic, typical Parkinson's disease (PD)
* At least 2 of 3 cardinal signs of PD
* Response to dopaminergic medication
* Mild cognitive impairment

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction within 6 months
* History of ventricular dysrhythmia requiring current therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Health education attention control
  Health education: Provision of general information about a variety of health topics
  Provision of general information about a variety of health
Period: Overall Study
Arm/Group | Physical Activity | Control
Started | 80 | 80
Completed | 59 | 59
Not Completed | 21 | 21
Not completed — Death | 7 | 11
Not completed — Lost to Follow-up | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity | Control | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.6) | 74.6 (8.3) | 74.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 78 | 80 | 158
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 80 | 160
Years of education [Mean (Standard Deviation); unit: years] | 13.6 (2.8) | 14.1 (2.5) | 13.8 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Cognitive Section of Alzheimer Disease Assessment Scale (ADAS-Cog) at Month 6
Description: The ADAS-Cog includes items assessing memory, orientation, language, and praxis. Scores range from 0-70 (higher scores indicate worse cognitive function). Change = Score at 6-month - Score at Baseline.
Time Frame: Baseline and 6 months
Population: number of participants analyzed: participants with ADAS-Cog scores at baseline and at 6 months. 4 participants in Physical Activity group and 6 participants in Control group did not have a score at 6 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Physical Activity | Control
Number analyzed (Participants) | 76 | 74
score on a scale | -0.24 (0.62) | 0.95 (0.78)
Statistical Analysis 1: Comparison: Physical Activity vs Control; Test type: Superiority; p = 0.2, Mixed Models Analysis; covariates: baseline age and years of education

2. Secondary Outcome: Change From Baseline on Cognitive Section of Alzheimer Disease Assessment Scale (ADAS-Cog) at Month 12
Description: The ADAS-Cog includes items assessing memory, orientation, language, and praxis. Scores range from 0-70 (higher scores indicate worse cognitive function). Change = Score at 12-month - Score at Baseline.
Time Frame: Baseline and 12 months
Population: number of participants analyzed: participants with ADAS-Cog scores at baseline and at 12 months. 17 participants in Physical Activity group and 15 participants in Control group did not have a score at 12 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physical Activity | Control
Number analyzed (Participants) | 63 | 65
units on a scale | 0.12 (0.79) | 2.60 (0.91)
Statistical Analysis 1: Comparison: Physical Activity vs Control; Test type: Superiority; p = 0.04, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline on Cognitive Section of Alzheimer Disease Assessment Scale (ADAS-Cog) at Month 18
Description: as for outcome 2
Time Frame: Baseline and 18 month
Population: number of participants analyzed: participants with ADAS-Cog scores at baseline and at 18 months. 21 participants in Physical Activity group and 21 participants in Control group did not have a score at 18 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Physical Activity | Control
Number analyzed (Participants) | 59 | 59
units on a scale | 0.40 (0.99) | 3.60 (1.03)
Statistical Analysis 1: Comparison: Physical Activity vs Control; Test type: Superiority; p = 0.02, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Physical Activity | Control
All-Cause Mortality (participants affected / at risk) | 7/80 | 11/80
Serious Adverse Events (participants affected / at risk) | 7/80 | 11/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=80) | Control (N=80)
Death (General disorders) | 7 (7) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT02248649/Prot_SAP_000.pdf